CLINICAL TRIAL: NCT06079554
Title: Microbiota and Metabolomics of Intestinal Type of Gastric Cancer in the Context of Atrophic Gastritis
Brief Title: Microbiota and Metabolomics of Intestinal Type of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Other Study IDs: 130027
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the gastric cancer group: 16 cases of intestinal type of gastric cancer under the background of atrophic gastritis
- the atrophic gastritis group: 16 cases of atrophic gastritis without gastric cancer matched according to gender, age, and degree of gastric atrophy

SUMMARY:
Compare with the gastric cavity without cancerous transformation in atrophic gastritis, analyze the microbiota and metabolomics changes in intestinal type of gastric cancer under the background of atrophic gastritis, and explore the relevant mechanisms.

DETAILED DESCRIPTION:
This study adopts a prospective cohort study. The expected recruitment time for all participants is 6 months, and all cases are cases who would receive magnifying endoscopy examination. The extent of atrophy and the presence of early gastric cancer are determined under magnifying endoscopy. Cases are chose into the gastric cancer group and atrophic gastritis group in a 1:1 ratio. There are 16 cases of intestinal type of gastric cancer under the background of atrophic gastritis, and 16 cases of atrophic gastritis without gastric cancer matched according to gender, age, and degree of gastric atrophy, totaling 32 cases. Analyze the characteristics of early gastric cancer under endoscopy, investigate the changes in microbiota and metabolomics of intestinal type of gastric cancer under the background of atrophic gastritis, and explore the relevant mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* •Intestinal type of gastric cancer or atrophic gastritis

  * Underwent Endoscopic submucosal dissection（ESD）

Exclusion Criteria:

* • have simultaneously other cancer

  * have severe systemic inflammatory disease ,serious illness such as diabetes, chronic lung diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We underwent magnifying staining endoscopy examination in our hospital and diagnosed cases of atrophic gastritis with or without gastric cancer under endoscopy.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Metabolomics results of lesions and atrophic gastritis. | 1year
  liquid chromatograph mass spectrometer metabolic profling

SECONDARY OUTCOMES:
microbiomics of lesions and atrophic gastritis. | 1 year
  16SrRNA analysis

OTHER OUTCOMES:
degree of gastric atrophy, | 1year
  According to the classification of Kimura-Takemoto Classification （C1-O3）
endoscopic observation | 1year
  NBI observation of atrophic background color, surrounding color of the lesion, lesion color, presence or absence of boundary transition zones, scattered intact glands within the lesion,presence of incomplete mesh patterns, and presence or absence of other early gastric cancer endoscopic manifestations.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No